CLINICAL TRIAL: NCT05878054
Title: The Hotspotters Project. Pursuing the Triple Aim in Hotspotters: Identification and Integrated Care
Brief Title: Pursuing the Triple Aim in Hotspotters: Identification and Integrated Care
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, rcvos, Associate Professor, Programma Manager Research, Leiden University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HTSPT
Record Dates: First submitted 2023-03-08; First posted 2023-05-26 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Complex Patient; Multimorbidity; Psychosocial Problem; Chronic Disease
Keywords: high care utilizer; complex patient; problems on multiple life domains; frequent flyer; hotspotter; high needs patient; integrated care; proactive care; personalised care; personalised care plan; positive health tool; multimorbidity; psychosocial problem
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Intervention Model Description: Stepped wedge cluster randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control period 2 months (Other): 2 months control period, followed by 12 months intervention, followed by 8 months observation
  Interventions: Other: Proactive, integrated and personalised care
- Control period 4 months (Other): 4 months control period, followed by 12 months intervention, followed by 6 months observation
  Interventions: Other: Proactive, integrated and personalised care
- Control period 6 months (Other): 6 months control period, followed by 12 months intervention, followed by 4 months observation
  Interventions: Other: Proactive, integrated and personalised care
- Control period 8 months (Other): 8 months control period, followed by 12 months intervention, followed by 2 months observation
  Interventions: Other: Proactive, integrated and personalised care

INTERVENTIONS:
Other: Proactive, integrated and personalised care — During the intervention patients receive proactive, integrated and personalised care. An intake consultation using Positive Health tool, or a similar method, the needs of each patient is assessed. In a multidisciplinary meeting with the GP, mental health care practice nurse, a social worker and the patient, a personalised care plan is made. The personal is executed and a care coordinator maintains proactive contact with the patient. Clinical follow-up will be done via a second multidisciplinary meeting.

SUMMARY:
Hotspotters are patients with complex care needs, defined by problems in multiple life domains and high acute care use. These patients often receive mismatched care, resulting in overuse of care and increased healthcare costs. Reliable data on (cost-)effective interventions for these patients are scarce. The goal of this study is to assess the cost-effectiveness of pro-active and integrated care. This approach includes: an intake consultation with Positive Health; multidisciplinary meetings with physician, mental healthcare nurse, social worker and the patient; a personalised care plan and proactive care management. We aim to include 200 patients, divided over 20 primary care practices.

DETAILED DESCRIPTION:
People with complex problems on multiple life domains, so called 'hotspotters', receive fragmented care. This is difficult to manage by patients and care providers , leading to little effect of care and persistent unmet needs. The accumulation and complexity of problems often leads to high medical expenses. Next to their high medical spending levels, hotspotters´ experiences with the healthcare system are low as the healthcare system is not (yet) successful in dealing with their needs. Interventions aimed at the complex situation of hotspotters in our current healthcare system might benefit by applying a Triple Aim approach. This approach aims to simultaneously improve the individual experience of care, reduce the cost of care per capita and improve the health of populations by offering proactive integrated care.

Is proactive integrated care costeffective and does it result in better patients experience than usual care after 12 months for patients with problems on multiple life domains? The intervention consists of: intake consultation assessing health on multiple domains using positive health or similar tool; multidisciplinary meetings with physician, mental healthcare nurse, social worker and patient, personalised care plan and proactive care management.

This stepped wedge cluster RCT aims to include 200 patients, divided over 20 primary care practices. All practices start with an observation period (2-8months), followed by the intervention (12 months) and follow-up (2-8months). Total duration of intervention is 22 months. We define Hotspotters as patients with at least two incidents of acute care utilisation (defined as out-of-office GP consultations, acute psychiatric care, emergency department visits and unplanned admissions) during the past year, and problems on two out of three health domains (chronic somatic, mental and/or social problems) based on diagnosis (coded with the International Classification of Primary Care) or medication (ATC) coding.

Primary outcome: Incremental cost-effectiveness from a societal perspective. Information on cost will be based on patient-reported data obtained by questionnaires supplied with data from the GP medical files (Huisarts informatie system, HIS) and CBSmicrodata. To assess the effectiveness the EQ-5D-5L will be used for determining quality of life.

Secondary outcomes: Insight into patients experience of care, quality of life, proactive coping, and self-efficacy. This information will be gathered using interviews, focus groups and questionnaires (SF-12, UPCC, PAM-13 and SE+IN itemlist). Process evaluation with the involved care professionals, integration level, the nature of the communication between healthcare provider and patient (HCCQ, OPTION5), and acceptability (AIM), appropriateness (IAM), feasibility (FIM) ,and perceived and experienced effectiveness of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* The patients are ≥ 18yrs
* The patients are registered within one of the participating GP practices.
* Patients with at least two acute care encounters in the past 12 months. Acute care encounter is defined as an encounter with out-of-hours GP service, emergency care or acute mental health care.Patients have problems registered in the GP Information system on at least two out of three of the following domains: somatic, mental or social. Somatic problems is having at least one ICPC code on the problem list. Mental problems is having at least one ICPC code from the "P"-chapter on either the problem list, as a reason for encounter, and/or having medication prescribed related to mental health problems. Social problems is having at least one ICPC code from the "Z"-chapter or as reason for encounter, and/or having medication prescribed related to social problems.

Exclusion Criteria:

* The patient is terminal.
* The patient is living in a residential home.
* The patient has dementia or a disability that prevents them from communicating effectively.The patient already has experience with the positive health tool.
* The patient is not competent to make decisions concerning their health. This wil be assessed by the patient's own general practitioner.
* Veto of the GP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Costs of care | 22 months
  Costs of care from a societal perspective is the summ of costs of care and loss of productivity due to illness or disease.
  Data on frequency and type of care utilization is gathered from the GP medical file, supplied with questions on mental health care use and need for addiction care. Productivity loss is determined via questionnaire. This data will be translated into cost using standard cost prices from the Dutch guideline for economic evaluations.
  Cost of care, together with Quality of life, will be used to assess cost-effectiveness from a societal perspective.
Quality adjusted life years | 22 months
  QALY measured by recurring EQ-5D-5L. Quality of life, together with cost of care, will be used to assess cost-effectiveness from a societal perspective.

SECONDARY OUTCOMES:
Self-regulation: Patient activation measure (PAM-13) | 22 months
  Self-regulation consists of measures of proactive coping, patient activation, self-efficacy and intention.
  The first is the validated Patient activation Measure (PAM-13). Patient Activation Measure (PAM-13), a validated 13-item questionnaire, assesses self-reported knowledge, skills and confidence in health management on 4-point scales ranging from 1 (totally disagree) to 4 (totally agree).
Self-regulation: Utrechtse Proactive Coping Compentence scale (UPCC) | 22 months
  Self-regulation consists of measures of proactive coping, patient activation, self-efficacy and intention.
  The Utrecht Proactive Coping Competence scale (UPCC) is a validated 21-item questionnaire that measures self-rated competence on proactive coping with 4-point scales ranging from 1 (not good) to 4 (very good)
Self-regulation: self-efficacy and intention itemlist (SE+IN itemlist) | 22 months
  Self-regulation consists of measures of proactive coping, patient activation, self-efficacy and intention. The Self-efficacy and Intention itemlist, specifically created for this study, measures self-management, self-efficacy, the intention to perform certain self-management behaviors and the presence of certain self-management behaviors.
  Action self-efficacy ("I am confident in my abilities to [ …] " and maintenance self-efficacy ("I am confident in my abilities to [….] when encountering obstacles") will be assessed in the Self-efficacy and Intention(SE+IN) itemlist for 8 items using 5-point scales, ranging from 1 (totally disagree) to 5 (totally agree). This addresses four key behaviours selected for the purpose of this study (adequate selfcare, maintaining daily structure, discussing concerns with care professionals, asking for help in a timely manner). Behavioural execution and intention to perform will also be assessed for each behaviour.
Experience of care: Healthcare climate questionnaire (HCCQ) | 22 months
  Experience of care: using measures of patient satisfaction, autonomy-supportive care and qualitative evaluation
  Researchers evaluate patients experiences with the personalised, integrated and proactive care approach using questionaires (HCCQ and mNPS, administerd 6 months after intervention start) and a qualitative approach (after intervention ends). The Health Care Climate Questionnaire (HCCQ) is a questionnaire on perceived degree of autonomy. It consists of 6-items, scored using 7-point likert scales. A higher score means that patients perceive a higher degree of autonomy.
Experience of care: modified Net Promotor scale (mNPS) | 22 months
  Experience of care: using measures of patient satisfaction, autonomy-supportive care and qualitative evaluation
  Researchers evaluate patients experiences with the personalised, integrated and proactive care approach using questionaires (HCCQ and mNPS, administerd 6 months after intervention start) and a qualitative approach (after intervention ends). The modified Net Promotor Scale (mNPS) consists of 2 patient-satisfaction-related items that are each scored between 0 and 10. A higher score means a higher satisfaction with the care received.
Experience of care: qualitative assessment | 22 months
  Experience of care uses measures of patient satisfaction, autonomy-supportive care and qualitative evaluation.
  Researchers evaluate patients experiences with the personalised, integrated and proactive care approach with both questionaires and a qualitative by means of a focus group. After the intervention, a focusgroup is organised to gather insight into the experiences of patients.
Administering of Positive Health methodology | 22 months
  the intake consultation and the first multidisciplinary meeting will be audio recorded to allow qualitative analysis of positive health methodology use. Themes, conversation techniques and the positive health topics addressed will be evaluated. Both deductive and inductive analyses will be employed to assess the use of positive health methodology, the importance of discussed life domains, patients' needs, problems and wishes, and how the personalised care plan was formed.
Health-related quality of life: short-form 12 health survey | 22 months
  Quality of life will also be assessed using the validated SF-12(12-items), including 8 dimensions, namely: bodily, pain, vitality (energy and fatigue), general mental health (psychological distress and well-being), general health perceptions, limitations in physical activities because of health problems, limitations in social activities because of physical or emotional problems, limitations in usual role activities because of emotional problems, and limitations in usual role activities because of physical health problems. Items are scored on a 3- or 5-points likert scale. The total SF=12 score ranges from 12 to 56 and a lower score means a better outcome.
  This questionnaire is administered thrice: at the start and end of intervention, and two months after ending the intervention.
Acceptability of Intervention Measure (AIM) | 22 months
  Acceptability, appropriateness, and feasibility will be measured using the The Acceptability of Intervention Measure (AIM). This will be done before the intervention starts and right after the intervention for each group of GP's. This information will be gathered from care professionals from participating as well as non-participating practices.
Level of shared decision making | 22 months
  Level of shared decision making will be based on audio recordings which will be scored by two independent observers using the validated OPTION5 questionnaire. If a participant is not comfortable with these recordings, the recordings may be skipped without further consequence for study participation.
Intervention Appropriateness Measure (IAM) | 22 months
  Intervention Appropriateness Measure (IAM), together with Feasibility of Intervention Measure (FIM), measures implementation outcomes that are often considered "leading indicators" of implementation success. This will be done before the intervention starts and right after the intervention for each group of GP's. This information will be gathered from care professionals from participating as well as non-participating practices.
Feasibility of Intervention Measure (FIM) | 22 months
  Feasibility of Intervention Measure (FIM), together with Intervention Appropriateness Measure (IAM), measures implementation outcomes that are often considered "leading indicators" of implementation success. This information will be gathered from care professionals from participating as well as non-participating practices.
Level of care integration | 22 months
  Professionals fill in the integrationmeter at the start and end of the intervention, resulting in a degree of care integration
Process evaluation following RE-AIM framework: reach, effectiveness, adoption, implementation and maintenance | 22 months
  Data on recruitment and population reach will be gathered during participant inclusion. Process evaluation of the study will be done simultaneous following the RE-AIM framework, thus providing insight on practicalities for future implementation. The five steps of the RE-AIM framework are:
  * Reach of target population: the number, proportion and representativeness of participants included in the study.
  * Effectiveness (or efficacy): the impact of the Hotspotters intervention is assessed in the primary outcome.
  * Adoption: The number, proportion and representativeness of care providers (that partook in the study) that is willing to initiate or continue the intervention outside of the study-context.
  * Implementation: the level of fidelity to intervention protocol per GP practice.
  * Maintenance: The extend in which the intervention becomes part of the routine care practice.

CONTACTS AND LOCATIONS:
Overall Officials: Rimke Vos, dr, Principal Investigator — Leiden University medical centre, health campus The Hague; Marc Bruijnzeels, dr, Principal Investigator — Leiden University medical centre, health campus The Hague
Locations (1):
- Leiden University Medical centre, department of Public Healht and Primary care (PHEG), location Health Campus The Hague, Leiden, Netherlands

REFERENCES:
- [Derived] Tiemes V, Leming KA, Borgdorff H, Bruijnzeels MA, van Gestel LC, Adriaanse MA, van der Wel M, van den Akker-van Marle EM, Numans ME, Vos RC. Hotspotters Project: a study protocol for a stepped wedge cluster RCT on the cost-effectiveness of 12-month proactive, integrated and personalised care for patients with problems on multiple life domains and high acute care use. BMJ Open. 2025 Aug 10;15(8):e087940. doi: 10.1136/bmjopen-2024-087940. PMID 40784776

DOCUMENTS (1):
  • Study Protocol (2023-04-24): https://cdn.clinicaltrials.gov/large-docs/54/NCT05878054/Prot_000.pdf